CLINICAL TRIAL: NCT01601002
Title: Does LEPR Polymorphism Predict Variability in Weight Gain Induced by Mirtazapine in the Treatment of Late Life Depression?
Brief Title: LEPR Polymorphism Weight Gain by Mirtazapine in Late Life Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Akshya Vasudev, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HSREB-102574
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Major Depressive Disorder
Keywords: Mirtazapine
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mirtazapine (Experimental): Mirtazapine in dosage of 7.5 mg to 45 mg/day
  Interventions: Drug: Mirtazapine

INTERVENTIONS:
Drug: Mirtazapine — Mirtazapine 7.5 to 45 mg/day, once daily, 12 weeks open label
  Other Names: Remeron

SUMMARY:
Patients with an episode of depression in late life prescribed mirtazapine recruited from a clinical sample will be monitored for weight and receive a blood test during their usual course of treatment to determine polymorphisms in a specific gene (LEPR) thought to affect weight gain.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 50 years
* meeting criteria for a diagnosis of major depressive disorder (DSM IV code 296.2x or 296.3x) as confirmed by a score > 20 on the HAM-D 24 items scale and a structured clinical interview using the SCID by a consultant psychiatrist

Exclusion Criteria:

* Treatment resistant depression (as defined by failure to respond to ≥2 adequate antidepressant trials)
* Major depressive disorder with psychosis (296.x4)
* Those with depression who fulfill the chronic specifier (MDE for >2 years)
* Significant Axis II pathology
* Previous trial with mirtazapine
* Concurrent antipsychotic usage
* Comorbid dementia (as confirmed by MMSE < 24)
* Substance misuse including drug and/or alcohol dependence/abuse in the past 3 months
* Bipolar disorder
* Schizophrenia
* Obsessive compulsive disorder
* Post traumatic stress disorder
* Eating disorder
* Head injury
* Recent stroke (< 3 months)
* Recent MI (< 3 months)
* Currently actively participating in structured/formal psychotherapy
* Being non ambulatory
* Those actively suicidal
* Those incapable of informed consent

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-06; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
increase in weight as measured in the clinic | Weeks 1,2,4,8 and 12 weeks

SECONDARY OUTCOMES:
Proportion of population achieving clinical response as measured by rate of fall in HAM-D 24 item scores | Start to end of study (12 weeks)
Proportion of patients achieving remission at end of study on HAM-D 24 (<11) | Start to end of study (12 weeks)
Frequency of adverse events | Start to end of study (12 weeks)
Percentage adhering to medication | Start to end of study (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Akshya Vasudev, MBBS, MD, MRCPsych, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada